CLINICAL TRIAL: NCT03010735
Title: Effects of Probiotics on Metabolism of Uremic Toxin in Patients With End Stage Renal Disease (ESRD)
Brief Title: Effects of Probiotics on the Patients With End Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: China Agricultural University (Other)
Collaborators: Peking University Aerospace Center Hospital (Other); General Hospital of Chinese Armed Police Forces (Other); Beijing Anzhen Hospital (Other); Beijing Biostats Technology Co. Ltd. (Unknown); Beijing Heyiyuan Biotech Co. Ltd. (Other)
Responsible Party: Principal Investigator, Fazheng Ren, Professor, China Agricultural University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAUPCKD-02
Record Dates: First submitted 2016-12-28; First posted 2017-01-05 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Kidney Failure, Chronic
Keywords: Kidney Failure, Chronic; Probiotics; Uremic toxins; Gastrointestinal Microbiome
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics (Active Comparator): The patient take two chewing tablet per day, which contain 4.0E+10 CFU of probiotics.
  Interventions: Dietary Supplement: probiotics
- Placebo (Placebo Comparator): The patient take two placebo chewing tablet per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: probiotics — Daily take 4.0E+10 CFU of probiotics
  Arms: Probiotics
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of oral administration of probiotics on the metabolism of uremic toxins, in the patients with End Stage Renal Disease (ESRD). One hundred and fifty hemodialysis patients are recruited, and a Double Blind Randomized Parallel Controlled Trial was performed.The microbiota-derived uremic toxin, such as indoxyl sulfate and p-cresol sulfate, are measured as Primary Outcome. The Fecal microbiome, fecal metabolites, blood metabolites, defecation, Gastrointestinal Symptoms The Kidney Disease Quality of Life and The Occurrence of Cardiovascular Event are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Patients who diagnosed as ESRD with hemodialysis
* Fixed hemodialysis cycle (average 3 times a week)
* Agree to take the products to be studied during the study period, and no longer take other fermented dairy products (live lactic acid bacteria drinks, cheese, yogurt, probiotic products, etc.)
* Agree to sign the informed consent form

Exclusion Criteria:

* Taking antibiotics or antifungal drugs within 30 days before the study
* Have serious allergic reaction to skim milk powder
* Researcher are not sure whether the subjects are willing or able to complete the study
* Subject participated in other research projects within two months before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in Microbiota-derived uremic toxin | 6 months
  follow up the patients at Month 0, 3, 6

SECONDARY OUTCOMES:
Changes in Fecal Microbiome | 6 months
  follow up the patients at Month 0, 3, 6
Changes in Fecal metabolites | 6 months
  follow up the patients at Month 0, 3, 6
Changes in Blood metabolites | 6 months
  follow up the patients at Month 0, 3, 6
Defecation questionnaire | 6 months
  follow up the patients at Month 0, 3, 6
Gastrointestinal Symptoms | 6 months
  follow up the patients at Month 0, 3, 6
The Kidney Disease Quality of Life | 6 months
  follow up the patients at Month 0, 3, 6
The Occurrence of Cardiovascular Event | 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fazheng Ren, PhD, Principal Investigator — China Agricultural Universtiy
Locations (3):
- China (3):
  - Beijing Anzhen Hospital, Beijing
  - General Hospital of Chinese Armed Police Forces, Beijing
  - Peking University Aerospace Centre Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaziri ND, Wong J, Pahl M, Piceno YM, Yuan J, DeSantis TZ, Ni Z, Nguyen TH, Andersen GL. Chronic kidney disease alters intestinal microbial flora. Kidney Int. 2013 Feb;83(2):308-15. doi: 10.1038/ki.2012.345. Epub 2012 Sep 19. PMID 22992469
- [Background] Poesen R, Windey K, Neven E, Kuypers D, De Preter V, Augustijns P, D'Haese P, Evenepoel P, Verbeke K, Meijers B. The Influence of CKD on Colonic Microbial Metabolism. J Am Soc Nephrol. 2016 May;27(5):1389-99. doi: 10.1681/ASN.2015030279. Epub 2015 Sep 23. PMID 26400570
- [Background] Koppe L, Mafra D, Fouque D. Probiotics and chronic kidney disease. Kidney Int. 2015 Nov;88(5):958-66. doi: 10.1038/ki.2015.255. Epub 2015 Sep 16. PMID 26376131
- [Background] Anders HJ, Andersen K, Stecher B. The intestinal microbiota, a leaky gut, and abnormal immunity in kidney disease. Kidney Int. 2013 Jun;83(6):1010-6. doi: 10.1038/ki.2012.440. Epub 2013 Jan 16. PMID 23325079
- [Background] Ramezani A, Raj DS. The gut microbiome, kidney disease, and targeted interventions. J Am Soc Nephrol. 2014 Apr;25(4):657-70. doi: 10.1681/ASN.2013080905. Epub 2013 Nov 14. PMID 24231662
- [Background] Poesen R, Claes K, Evenepoel P, de Loor H, Augustijns P, Kuypers D, Meijers B. Microbiota-Derived Phenylacetylglutamine Associates with Overall Mortality and Cardiovascular Disease in Patients with CKD. J Am Soc Nephrol. 2016 Nov;27(11):3479-3487. doi: 10.1681/ASN.2015121302. Epub 2016 May 26. PMID 27230658
- [Background] Meyer TW, Hostetter TH. Uremia. N Engl J Med. 2007 Sep 27;357(13):1316-25. doi: 10.1056/NEJMra071313. No abstract available. PMID 17898101
- [Background] Aronov PA, Luo FJ, Plummer NS, Quan Z, Holmes S, Hostetter TH, Meyer TW. Colonic contribution to uremic solutes. J Am Soc Nephrol. 2011 Sep;22(9):1769-76. doi: 10.1681/ASN.2010121220. Epub 2011 Jul 22. PMID 21784895